CLINICAL TRIAL: NCT04239872
Title: Optimizing Fluoride Retention in the Mouth of Older Adults With Distinct Salivary Flow Rates
Brief Title: Fluoride Retention in the Mouth of Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Livia Tenuta, DDS, MS, PhD, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HUM00159624; UL1TR002240 (NIH)
Record Dates: First submitted 2020-01-15; First posted 2020-01-27 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Hyposalivation
MeSH Terms: conditions — Xerostomia | interventions — Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluoride mouthwash alone, then Calcium mouthwash before a fluoride mouthwash (Experimental): Participants with normal to dry mouth will first test a Fluoride mouthwash containing 226 ppm of fluoride, and fluoride concentration in saliva and dental biofilm will be assessed overtime for up to 2 hours. After a washout period of at least 3 days, they will then test a Calcium mouthwash (150 milimolars of calcium) immediately before the Fluoride mouthwash, and fluoride concentration in saliva and dental biofilm will be assessed overtime for up to 2 hours.
  Interventions: Drug: Fluoride mouthwash; Drug: Calcium and fluoride mouthwash
- Calcium mouthwash before a fluoride mouthwash, then Fluoride mouthwash alone (Experimental): Participants with normal to dry mouth will first test a Calcium mouthwash (150 milimolars of calcium) immediately before a Fluoride mouthwash containing 226 ppm of fluoride, and fluoride concentration in saliva and dental biofilm will be assessed overtime for up to 2 hours. After a washout period of at least 3 days, they will then test the Fluoride mouthwash alone, and fluoride concentration in saliva and dental biofilm will be assessed overtime for up to 2 hours.
  Interventions: Drug: Fluoride mouthwash; Drug: Calcium and fluoride mouthwash

INTERVENTIONS:
Drug: Fluoride mouthwash — Sodium fluoride, at a concentration of 0.05% (226 parts per million (ppm) of fluoride), will be used to rinse the mouth for 1 minute and expectorated.
  Other Names: Fluoride rinse
Drug: Calcium and fluoride mouthwash — Calcium lactate, at a concentration of 150 milimolar, will be used to rinse the mouth for 1 minute and expectorated; immediately after, a sodium fluoride rinse, at a concentration of 0.05% (226 ppm of fluoride), will be used to rinse the mouth for 1 minute, and expectorated.
  Other Names: Calcium and fluoride rinse

SUMMARY:
Individuals with dry mouth (a reduction in the production of saliva) suffer from high rates of oral diseases. Dry mouth is a common problem among older individuals, because many medications to control chronic conditions (such as blood pressure, bladder-control problems and depression) reduce the flow of saliva. For these individuals, fluoride is used to maintain a good oral health. Usually, higher fluoride concentration products, such as prescription toothpastes, are recommended. In this project, the ability to increase fluoride retention in the mouth by using calcium before a conventional fluoride rinse will be tested in older adults with a range of salivary flow rates. This approach was never tested in patients with dry mouth, for whom the treatment with calcium may also be beneficial. A crossover, clinical study with two experimental phases will be conducted, in which patients with a range of saliva flows (from normal to dry mouth) will rinse with a fluoride rinse only (used at over the counter concentration), or a fluoride rinse preceded by a calcium rinse. The concentration of fluoride and calcium in the saliva and dental plaque residues will be determined up to two hours after the rinse(s), to test the effect of the approach to optimize fluoride retention in the mouth of patients with dry mouth.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Good general health as evidenced by medical history
* Good oral health as evidenced by a clinical oral exam
* Having at least 20 teeth in the mouth, being at least 4 (natural or crowned) teeth in all four quadrants of the mouth
* Having salivary flow rate ranging from normal to hyposalivation according to direct flow rate determination methods
* Agreement to adhere to the study protocol

Exclusion Criteria:

* Unable to understand and/or follow study instructions
* Active periodontitis
* Oral pain
* In need of urgent dental care

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Livia M Tenuta, DDS, MS, PhD, Principal Investigator — Associate Professor, University of Michigan
Locations (1):
- School of Dentistry, University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluoride Mouthwash Alone, Then Calcium Mouthwash Before a Fluoride Mouthwash: Participants with normal to dry mouth first tested a Fluoride mouthwash containing 226 ppm of fluoride, and fluoride concentration in saliva and dental biofilm was assessed overtime for up to 2 hours. After a washout period of at least 3 days, they then tested a Calcium mouthwash (150 millimoles per liter of calcium) immediately before the Fluoride mouthwash, and fluoride concentration in saliva and dental biofilm was assessed overtime for up to 2 hours.
- Calcium Mouthwash Before a Fluoride Mouthwash, Then Fluoride Mouthwash Alone: Participants with normal to dry mouth first tested a Calcium mouthwash (150 millimoles per liter of calcium) immediately before a Fluoride mouthwash containing 226 ppm of fluoride, and fluoride concentration in saliva and dental biofilm was assessed overtime for up to 2 hours. After a washout period of at least 3 days, they then tested the Fluoride mouthwash alone, and fluoride concentration in saliva and dental biofilm was assessed overtime for up to 2 hours.
Period: Overall Study
Arm/Group | Fluoride Mouthwash Alone, Then Calcium Mouthwash Before a Fluoride Mouthwash | Calcium Mouthwash Before a Fluoride Mouthwash, Then Fluoride Mouthwash Alone
Started | 11 | 9
Completed | 11 | 8
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants With Normal Salivary Flow to Dry Mouth: Participants were randomly assigned to two arms, with varying sequence of treatment used, under a crossover design: Fluoride mouthwash alone, then Calcium mouthwash before a fluoride mouthwash; OR Calcium mouthwash before a fluoride mouthwash, then Fluoride mouthwash alone
  Fluoride mouthwash consisted of Sodium fluoride, at a concentration of 0.05% (226 parts per million (ppm) of fluoride), used to rinse the mouth for 1 minute and expectorated.
  Calcium and fluoride mouthwash: Calcium lactate, at a concentration of 150 millimoles per liter, used to rinse the mouth for 1 minute and expectorated; immediately after, a sodium fluoride rinse, at a concentration of 0.05% (226 ppm of fluoride), used to rinse the mouth for 1 minute, and expectorated.
Arm/Group | Participants With Normal Salivary Flow to Dry Mouth
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20
Unstimulated salivary flow rate, mL/min [Mean (Standard Deviation); unit: mL/min] | 0.3 (0.33)
Stimulated salivary flow rate, mL/min [Mean (Standard Deviation); unit: mL/min] | 1.21 (0.87)

OUTCOME MEASURES:

1. Primary Outcome: Fluoride Concentration in Dental Biofilm Fluid at Baseline
Description: Dental biofilm was collected at baseline (before mouthwash(es)), and the fluid phase was separated using centrifugation. Fluoride concentration in the dental biofilm fluid was measured using an ion-specific electrode adapted for microanalysis.
Time Frame: Baseline
Population: A smaller number of participants analyzed for this variable means that they did not have sample collected at this time point, or that the amount collected was not enough for the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: parts per million (ppm) of fluoride
Groups:
- Fluoride Mouthwash: Participants with normal salivary flow to dry mouth were treated, in a crossover design, with two interventions: a fluoride mouthwash alone, or a fluoride mouthwash preceded by a calcium mouthwash.
  Participants were randomized to determine which intervention they used in the first experimental phase; the other intervention will the tested in the second phase.
  This arm refers to the use of the fluoride mouthwash: Sodium fluoride, at a concentration of 0.05% (226 parts per million (ppm) of fluoride), was used to rinse the mouth for 1 minute and expectorated.
- Calcium Mouthwash Before Fluoride Mouthwash: Participants with normal salivary flow to dry mouth were treated, in a crossover design, with two interventions: a fluoride mouthwash alone, or a fluoride mouthwash preceded by a calcium mouthwash.
  Participants were randomized to determine which intervention they used in the first experimental phase; the other intervention will the tested in the second phase.
  This arm refers to the use of the calcium mouthwash before the fluoride mouthwash: Calcium lactate, at a concentration of 150 millimolar, was used to rinse the mouth for 1 minute and expectorated; immediately after, a sodium fluoride rinse, at a concentration of 0.05% (226 ppm of fluoride), was used to rinse the mouth for 1 minute, and expectorated.
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 14 | 13
parts per million (ppm) of fluoride | 0.24 [0.18 to 0.32] | 0.22 [0.17 to 0.29]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; A paired t-test was used to compare the two groups. To obtain normal distribution, data used in the statistical analysis were transformed to the log10; Test type: Superiority; p = 0.8412, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 11 pairs of data, DF=10; Mean Difference (Net) = -0.00778, 95% CI 2-sided [-0.09209 to 0.07653] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

2. Primary Outcome: Fluoride Concentration in Dental Biofilm Fluid at 15 Minutes
Description: Dental biofilm was collected 15 minutes after mouthwash(es), and the fluid phase was separated using centrifugation. Fluoride concentration in the dental biofilm fluid was measured using an ion-specific electrode adapted for microanalysis.
Time Frame: 15 minutes after mouthwash(es)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: parts per million (ppm) of fluoride
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 14 | 14
parts per million (ppm) of fluoride | 15.27 [7.84 to 29.76] | 12.29 [9.46 to 15.98]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6504, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 12 pairs of data, DF=11; Mean Difference (Net) = -0.06907, 95% CI 2-sided [-0.3955 to 0.2573] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

3. Primary Outcome: Fluoride Concentration in Dental Biofilm Fluid at 60 Minutes
Description: Dental biofilm was collected 60 minutes after mouthwash(es), and the fluid phase was separated using centrifugation. Fluoride concentration in the dental biofilm fluid was measured using an ion-specific electrode adapted for microanalysis.
Time Frame: 60 minutes after mouthwash(es)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: parts per million (ppm) of fluoride
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 13 | 15
parts per million (ppm) of fluoride | 1.57 [0.79 to 3.11] | 4.07 [2.63 to 6.31]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0024, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 11 pairs of data, DF=10; Mean Difference (Net) = 0.5307, 95% CI 2-sided [0.2372 to 0.8243] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

4. Primary Outcome: Fluoride Concentration in Dental Biofilm Fluid at 120 Minutes
Description: Dental biofilm was collected 120 minutes after mouthwash(es), and the fluid phase was separated using centrifugation. Fluoride concentration in the dental biofilm fluid was measured using an ion-specific electrode adapted for microanalysis.
Time Frame: 120 minutes after mouthwash(es)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: parts per million (ppm) of fluoride
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 16 | 10
parts per million (ppm) of fluoride | 0.63 [0.40 to 0.99] | 2.58 [1.33 to 5.00]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0013, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 9 pairs of data, DF=8; Mean Difference (Net) = 0.5643, 95% CI 2-sided [0.2938 to 0.8348] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

5. Primary Outcome: Fluoride Concentration in Dental Biofilm Solids at Baseline
Description: Dental biofilm was collected at baseline (before mouthwash(es)). The fluid phase of the biofilm was collected after centrifugation, and the remaining solids were treated with strong acid for dissolution of fluoride reservoirs. Solids remaining after acid extraction were treated with strong alkali for total dissolution of the biofilm and estimation of biofilm mass by protein concentration. Fluoride concentration in the dental biofilm solids acid extract was measured using an ion-specific electrode adapted for microanalysis; protein concentration in the alkali extract was determined using the Lowry colorimetric method. Fluoride concentration in the biofilm was expressed as micrograms of fluoride/milligrams of protein.
Time Frame: Baseline
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms fluoride/milligram protein
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 17 | 16
micrograms fluoride/milligram protein | 0.17 [0.09 to 0.32] | 0.13 [0.07 to 0.24]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2041, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 15 pairs of data, DF=14; Mean Difference (Net) = -0.1135, 95% CI 2-sided [-0.2964 to 0.06929] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

6. Primary Outcome: Fluoride Concentration in Dental Biofilm Solids at 15 Minutes
Description: Dental biofilm was collected 15 minutes after mouthwash(es). The fluid phase of the biofilm was collected after centrifugation, and the remaining solids were treated with strong acid for dissolution of fluoride reservoirs. Solids remaining after acid extraction were treated with strong alkali for total dissolution of the biofilm and estimation of biofilm mass by protein concentration. Fluoride concentration in the dental biofilm solids acid extract was measured using an ion-specific electrode adapted for microanalysis; protein concentration in the alkali extract was determined using the Lowry colorimetric method. Fluoride concentration in the biofilm was expressed as micrograms of fluoride/milligrams of protein.
Time Frame: 15 minutes after mouthwash(es)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms fluoride/milligram protein
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 16 | 14
micrograms fluoride/milligram protein | 0.44 [0.27 to 0.73] | 5.30 [3.87 to 7.27]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 13 pairs of data, DF=12; Mean Difference (Net) = 1.095, 95% CI 2-sided [0.7736 to 1.416] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

7. Primary Outcome: Fluoride Concentration in Dental Biofilm Solids at 60 Minutes
Description: Dental biofilm will be collected 60 minutes after mouthwash(es). The fluid phase of the biofilm was collected after centrifugation, and the remaining solids were treated with strong acid for dissolution of fluoride reservoirs. Solids remaining after acid extraction were treated with strong alkali for total dissolution of the biofilm and estimation of biofilm mass by protein concentration. Fluoride concentration in the dental biofilm solids acid extract was measured using an ion-specific electrode adapted for microanalysis; protein concentration in the alkali extract was determined using the Lowry colorimetric method. Fluoride concentration in the biofilm was expressed as micrograms of fluoride/milligrams of protein.
Time Frame: 60 minutes after mouthwash(es)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms fluoride/miligram protein
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 15 | 16
micrograms fluoride/miligram protein | 0.23 [0.10 to 0.53] | 5.98 [4.36 to 8.21]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 13 pairs of data, DF=12; Mean Difference (Net) = 1.469, 95% CI 2-sided [1.112 to 1.825] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

8. Primary Outcome: Fluoride Concentration in Dental Biofilm Solids at 120 Minutes
Description: Dental biofilm was collected 120 minutes after mouthwash(es). The fluid phase of the biofilm was collected after centrifugation, and the remaining solids were treated with strong acid for dissolution of fluoride reservoirs. Solids remaining after acid extraction were treated with strong alkali for total dissolution of the biofilm and estimation of biofilm mass by protein concentration. Fluoride concentration in the dental biofilm solids acid extract was measured using an ion-specific electrode adapted for microanalysis; protein concentration in the alkali extract was determined using the Lowry colorimetric method. Fluoride concentration in the biofilm was expressed as micrograms of fluoride/milligrams of protein.
Time Frame: 120 minutes after mouthwash(es)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms fluoride/miligram protein
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 18 | 15
micrograms fluoride/miligram protein | 0.18 [0.08 to 0.40] | 4.84 [3.61 to 6.49]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 14 pairs of data, DF=13; Mean Difference (Net) = 1.549, 95% CI 2-sided [1.081 to 2.017] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

9. Primary Outcome: Area Under the Curve of Fluoride Concentration in Dental Biofilm Fluid Overtime
Description: Fluoride concentration in dental biofilm fluid collected at baseline (before mouthwash(es)), 15, 60 and 120 minutes after mouthwash(es) was expressed as the area under the curve of fluoride concentration in dental biofilm fluid as a function of time (parts per million x min).
Time Frame: Baseline, 15, 60 and 120 minutes after mouthwash(es)
Population: The area under the curve was calculated only for participants with all time points collected. This accounts for the smaller number of participants analyzed for this variable.
Measure: Mean (Standard Deviation); unit: parts per million x minutes
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 10 | 8
parts per million x minutes | 841.6 (543.2) | 764.4 (234.1)
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; A paired t-test was used to compare the two groups; Test type: Superiority; p = 0.5543, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 6 pairs of data, DF=5; Mean Difference (Net) = -115.6, 95% CI 2-sided [-584.8 to 353.6] — Treatment difference = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

10. Primary Outcome: Area Under the Curve of Fluoride Concentration in Dental Biofilm Solids Overtime
Description: Fluoride concentration in dental biofilm solids collected at baseline (before mouthwash(es)), 15, 60 and 120 minutes after mouthwash(es) was expressed as the area under the curve of fluoride concentration in dental biofilm solids as a function of time (micrograms of fluoride x minutes/ milligram of proteins).
Time Frame: Baseline, 15, 60 and 120 minutes after mouthwash
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: microgram fluoride/milligram prot x min
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 14 | 10
microgram fluoride/milligram prot x min | 37.85 [18.33 to 78.14] | 521.2 [376.7 to 721.2]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0003, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 8 pairs of data, DF=7; Mean Difference (Net) = 1.328, 95% CI 2-sided [0.8420 to 1.814] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

11. Secondary Outcome: Fluoride Concentration in Saliva at Baseline
Description: Unstimulated saliva was collected at baseline (before mouthwash(es)), for 5 minutes. Fluoride concentration in unstimulated saliva was measured using an ion-specific electrode adapted for microanalysis.
Time Frame: Baseline
Population: A smaller number of participants analyzed for this variable means that they did not have a sample collected at this time point, or that the amount collected was not enough for the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: parts per million (ppm) of fluoride
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 19 | 20
parts per million (ppm) of fluoride | 0.14 [0.09 to 0.21] | 0.11 [0.09 to 0.13]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2824, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 19 pairs of data, DF=18; Mean Difference (Net) = -0.09023, 95% CI 2-sided [-0.2613 to 0.08082] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

12. Secondary Outcome: Fluoride Concentration in Saliva at 16 Minutes
Description: Unstimulated saliva was collected 16 minutes after mouthwash(es), for 5 minutes. Fluoride concentration in unstimulated saliva was measured using an ion-specific electrode adapted for microanalysis.
Time Frame: 16-21 minutes after mouthwash(es)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: parts per million (ppm) of fluoride
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 17 | 20
parts per million (ppm) of fluoride | 4.60 [2.70 to 7.81] | 20.36 [15.08 to 27.48]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0002, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 17 pairs of data, DF=16; Mean Difference (Net) = 0.6269, 95% CI 2-sided [0.3488 to 0.9050] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

13. Secondary Outcome: Fluoride Concentration in Saliva at 30 Minutes
Description: Unstimulated saliva was collected 30 minutes after mouthwash(es), for 5 minutes. Fluoride concentration in unstimulated saliva was measured using an ion-specific electrode adapted for microanalysis.
Time Frame: 30-35 minutes after mouthwash(es)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: parts per million (ppm) of fluoride
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 17 | 18
parts per million (ppm) of fluoride | 2.18 [1.21 to 3.90] | 17.05 [14.54 to 19.99]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 17 pairs of data, DF=16; Mean Difference (Net) = 0.8946, 95% CI 2-sided [0.6671 to 1.122] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

14. Secondary Outcome: Fluoride Concentration in Saliva at 61 Minutes
Description: Unstimulated saliva was collected 61 minutes after mouthwash(es), for 5 minutes. Fluoride concentration in unstimulated saliva was measured using an ion-specific electrode adapted for microanalysis.
Time Frame: 61-66 minutes after mouthwash(es)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: parts per million (ppm) of fluoride
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 18 | 20
parts per million (ppm) of fluoride | 1.07 [0.67 to 1.72] | 9.98 [6.89 to 14.50]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 18 pairs of data, DF=17; Mean Difference (Net) = 0.9730, 95% CI 2-sided [0.7597 to 1.186] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

15. Secondary Outcome: Fluoride Concentration in Saliva at 90 Minutes
Description: Unstimulated saliva was collected 90 minutes after mouthwash(es), for 5 minutes. Fluoride concentration in unstimulated saliva was measured using an ion-specific electrode adapted for microanalysis.
Time Frame: 90-95 minutes after mouthwash(es)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: parts per million (ppm) of fluoride
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 18 | 19
parts per million (ppm) of fluoride | 0.80 [0.49 to 1.32] | 7.66 [5.61 to 10.5]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 18 pairs of data, DF=17; Mean Difference (Net) = 0.9827, 95% CI 2-sided [0.7758 to 1.19] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

16. Secondary Outcome: Fluoride Concentration in Saliva at 121 Minutes
Description: Unstimulated saliva was collected 121 minutes after mouthwash(es), for 5 minutes. Fluoride concentration in unstimulated saliva was measured using an ion-specific electrode adapted for microanalysis.
Time Frame: 121-126 minutes after mouthwash(es)
Measure: Geometric Mean (95% Confidence Interval); unit: parts per million (ppm) of fluoride
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 19 | 20
parts per million (ppm) of fluoride | 0.46 [0.30 to 0.69] | 3.71 [2.18 to 6.30]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 19 pairs of data, DF=18; Mean Difference (Net) = 0.9181, 95% CI 2-sided [0.6573 to 1.179] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

17. Secondary Outcome: Calcium Concentration in Dental Biofilm Fluid at Baseline
Description: Dental biofilm will be collected at baseline (before mouthwash(es)), and the fluid phase will be separated using centrifugation. Calcium concentration in the dental biofilm fluid will be measured using an ion-specific electrode adapted for microanalysis, and will be expressed in millimolar.
Time Frame: Baseline
Population: Due to the small amount of biofilm collected from participants, resulting in a reduced biofilm fluid volume, there was not enough sample left for calcium measurement after fluoride concentration in the fluid was determined.
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Calcium Concentration in Dental Biofilm Fluid at 15 Minutes
Description: Dental biofilm will be collected 15 minutes after mouthwash(es), and the fluid phase will be separated using centrifugation. Calcium concentration in the dental biofilm fluid will be measured using an ion-specific electrode adapted for microanalysis, and will be expressed in millimolar.
Time Frame: 15 minutes after mouthwash(es)
Population: as for outcome 17
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Calcium Concentration in Dental Biofilm Fluid at 60 Minutes
Description: Dental biofilm will be collected 60 minutes after mouthwash(es), and the fluid phase will be separated using centrifugation. Calcium concentration in the dental biofilm fluid will be measured using an ion-specific electrode adapted for microanalysis, and will be expressed in millimolar.
Time Frame: 60 minutes after mouthwash(es)
Population: as for outcome 17
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Calcium Concentration in Dental Biofilm Fluid at 120 Minutes
Description: Dental biofilm will be collected 120 minutes after mouthwash(es), and the fluid phase will be separated using centrifugation. Calcium concentration in the dental biofilm fluid will be measured using an ion-specific electrode adapted for microanalysis, and will be expressed in millimolar.
Time Frame: 120 minutes after mouthwash(es)
Population: as for outcome 17
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Calcium Concentration in Dental Biofilm Solids at Baseline
Description: Dental biofilm was collected at baseline (before mouthwash(es)). The fluid phase of the biofilm was collected after centrifugation, and the remaining solids were treated with strong acid for dissolution of calcium reservoirs. Solids remaining after acid extraction were treated with strong alkali for total dissolution of the biofilm and estimation of biofilm mass by protein concentration. Calcium concentration in the dental biofilm solids acid extract was measured using a colorimetric reaction (Arsenazo III); protein concentration in the alkali extract was determined using the Lowry colorimetric method. Calcium concentration in the biofilm was expressed as micrograms of calcium/milligrams of protein.
Time Frame: Baseline
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms calcium/miligram protein
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 17 | 16
micrograms calcium/miligram protein | 5.74 [3.78 to 8.72] | 4.67 [3.01 to 7.23]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3283, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 15 pairs of data, DF=14; Mean Difference (Net) = -0.05652, 95% CI 2-sided [-0.1762 to 0.06829] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

22. Secondary Outcome: Calcium Concentration in Dental Biofilm Solids at 15 Minutes
Description: Dental biofilm was collected 15 minutes after mouthwash(es). The fluid phase of the biofilm was collected after centrifugation, and the remaining solids were treated with strong acid for dissolution of calcium reservoirs. Solids remaining after acid extraction were treated with strong alkali for total dissolution of the biofilm and estimation of biofilm mass by protein concentration. Calcium concentration in the dental biofilm solids acid extract was measured using a colorimetric reaction (Arsenazo III); protein concentration in the alkali extract was determined using the Lowry colorimetric method. Calcium concentration in the biofilm was expressed as micrograms of calcium/milligrams of protein.
Time Frame: 15 minutes after mouthwash(es)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms calcium/miligram protein
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 16 | 14
micrograms calcium/miligram protein | 4.48 [3.02 to 6.65] | 8.88 [6.80 to 11.60]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0058, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 13 pairs of data, DF=12; Mean Difference (Net) = 0.3411, 95% CI 2-sided [0.1189 to 0.5633] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

23. Secondary Outcome: Calcium Concentration in Dental Biofilm Solids at 60 Minutes
Description: Dental biofilm was collected 60 minutes after mouthwash(es). The fluid phase of the biofilm was collected after centrifugation, and the remaining solids were treated with strong acid for dissolution of calcium reservoirs. Solids remaining after acid extraction were treated with strong alkali for total dissolution of the biofilm and estimation of biofilm mass by protein concentration. Calcium concentration in the dental biofilm solids acid extract was measured using a colorimetric reaction (Arsenazo III); protein concentration in the alkali extract was determined using the Lowry colorimetric method. Calcium concentration in the biofilm was expressed as micrograms of calcium/milligrams of protein.
Time Frame: 60 minutes after mouthwash(es)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms calcium/miligram protein
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 15 | 16
micrograms calcium/miligram protein | 6.64 [3.40 to 13.0] | 12.4 [8.22 to 18.8]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0213, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 13 pairs of data, DF=12; Mean Difference (Net) = 0.2976, 95% CI 2-sided [0.05266 to 0.5426] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

24. Secondary Outcome: Calcium Concentration in Dental Biofilm Solids at 120 Minutes
Description: Dental biofilm was collected 120 minutes after mouthwash(es). The fluid phase of the biofilm was collected after centrifugation, and the remaining solids were treated with strong acid for dissolution of calcium reservoirs. Solids remaining after acid extraction were treated with strong alkali for total dissolution of the biofilm and estimation of biofilm mass by protein concentration. Calcium concentration in the dental biofilm solids acid extract was measured using a colorimetric reaction (Arsenazo III); protein concentration in the alkali extract was determined using the Lowry colorimetric method. Calcium concentration in the biofilm was expressed as micrograms of calcium/milligrams of protein.
Time Frame: 120 minutes after mouthwash(es)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms calcium/miligram protein
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 18 | 15
micrograms calcium/miligram protein | 5.08 [2.94 to 8.77] | 9.66 [6.91 to 13.5]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.014, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 14 pairs of data, DF=13; Mean Difference (Net) = 0.3120, 95% CI 2-sided [0.07454 to 0.5495] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

25. Secondary Outcome: Calcium Concentration in Saliva at Baseline
Description: Unstimulated saliva was collected at baseline (before mouthwash(es)), for 5 minutes. Calcium concentration in unstimulated saliva was measured using a colorimetric reaction (Arsenazo III).
Time Frame: Baseline
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milimolar
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 17 | 19
milimolar | 1.57 (0.64) | 1.76 (0.64)
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; A paired t-test was used to compare the two groups; Test type: Superiority; p = 0.1393, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 17 pairs of data, DF=16; Mean Difference (Net) = 0.2524, 95% CI 2-sided [-0.09153 to 0.5962] — Treatment difference = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

26. Secondary Outcome: Calcium Concentration in Saliva at 16 Minutes
Description: Unstimulated saliva was collected at 16 minutes after mouthwash(es), for 5 minutes. Calcium concentration in unstimulated saliva was measured using a colorimetric reaction (Arsenazo III).
Time Frame: 16-21 minutes after mouthwash(es)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: milimolar
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 16 | 19
milimolar | 1.14 [0.92 to 1.42] | 2.38 [1.65 to 3.43]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0009, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 16 pairs of data, DF=15; Mean Difference (Net) = 0.2921, 95% CI 2-sided [0.1414 to 0.4427] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

27. Secondary Outcome: Calcium Concentration in Saliva at 30 Minutes
Description: Unstimulated saliva was collected at 30 minutes after mouthwash(es), for 5 minutes. Calcium concentration in unstimulated saliva was measured using a colorimetric reaction (Arsenazo III).
Time Frame: 30-35 minutes after mouthwash(es)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: milimolar
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 16 | 18
milimolar | 1.12 [0.87 to 1.45] | 2.03 [1.62 to 2.53]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0008, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 16 pairs of data, DF=15; Mean Difference (Net) = 0.2433, 95% CI 2-sided [0.1195 to 0.3671] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

28. Secondary Outcome: Calcium Concentration in Saliva at 61 Minutes
Description: Unstimulated saliva was collected at 61 minutes after mouthwash(es), for 5 minutes. Calcium concentration in unstimulated saliva was measured using a colorimetric reaction (Arsenazo III).
Time Frame: 61-66 minutes after mouthwash(es)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milimolar
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 18 | 17
milimolar | 1.62 (0.60) | 2.01 (0.60)
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; A paired t-test was used to compare the two groups; Test type: Superiority; p = 0.1515, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 16 pairs of data, DF=15; Mean Difference (Net) = 0.3306, 95% CI 2-sided [-0.1356 to 0.7969] — Treatment difference = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

29. Secondary Outcome: Calcium Concentration in Saliva at 90 Minutes
Description: Unstimulated saliva was collected at 90 minutes after mouthwash(es), for 5 minutes. Calcium concentration in unstimulated saliva was measured using a colorimetric reaction (Arsenazo III).
Time Frame: 90-95 minutes after mouthwash(es)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: milimolar
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 17 | 19
milimolar | 1.50 [1.21 to 1.88] | 1.74 [1.47 to 2.07]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1712, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 17 pairs of data, DF=16; Mean Difference (Net) = 0.04851, 95% CI 2-sided [-0.02327 to 0.1203] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

30. Secondary Outcome: Calcium Concentration in Saliva at 121 Minutes
Description: Unstimulated saliva was collected at 121 minutes after mouthwash(es), for 5 minutes. Calcium concentration in unstimulated saliva was measured using a colorimetric reaction (Arsenazo III).
Time Frame: 121-126 minutes after mouthwash(es)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milimolar
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 19 | 19
milimolar | 1.60 (0.57) | 1.80 (0.59)
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; A paired t-test was used to compare the two groups; Test type: Superiority; p = 0.1188, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 18 pairs of data, DF=17; Mean Difference (Net) = 0.2789, 95% CI 2-sided [-0.07934 to 0.6371] — Treatment difference = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

31. Secondary Outcome: Area Under the Curve of Fluoride Concentration in Saliva Overtime
Description: Fluoride concentration in unstimulated saliva collected at baseline (before mouthwash(es)), 16, 30, 61, 90 and 121 minutes after mouthwash(es) was expressed as the area under the curve of fluoride concentration in saliva as a function of time.
Time Frame: Baseline, 16, 30, 61, 90 and 121 minutes after mouthwash(es)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: parts per million x minutes
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 14 | 18
parts per million x minutes | 186 [111 to 312] | 1415 [1170 to 1713]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 14 pairs of data, DF=13; Mean Difference (Net) = 0.8956, 95% CI 2-sided [0.7205 to 1.071] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

32. Secondary Outcome: Area Under the Curve of Calcium Concentration in Dental Biofilm Fluid Overtime
Description: Calcium concentration in dental biofilm fluid collected at baseline (before mouthwash(es)), 15, 60 and 120 minutes after mouthwash(es) will be expressed as the area under the curve of calcium concentration in dental biofilm fluid as a function of time (millimolar x min).
Time Frame: Baseline, 15, 60 and 120 minutes after mouthwash(es)
Population: Due to the small amount of biofilm collected from participants, resulting in a reduced biofilm fluid volume, there was not enough sample left for calcium measurement after fluoride concentration in the fluid was determined. Therefore, the area under the curve could not be estimated for this variable.
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Area Under the Curve of Calcium Concentration in Dental Biofilm Solids Overtime
Description: Calcium concentration in dental biofilm solids collected at baseline (before mouthwash(es)), 15, 60 and 120 minutes after mouthwash(es) was expressed as the area under the curve of calcium concentration in dental biofilm solids as a function of time.
Time Frame: Baseline, 15, 60 and 120 minutes after mouthwash(es)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms calcium x time/milligram prot
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 14 | 10
micrograms calcium x time/milligram prot | 780 [424 to 1436] | 1165 [732 to 1854]
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0475, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 8 pairs of data, DF=7; Mean Difference (Net) = 0.3199, 95% CI 2-sided [0.004686 to 0.6351] — Treatment difference of transformed (log10) data = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

34. Secondary Outcome: Area Under the Curve of Calcium Concentration in Saliva Overtime
Description: Calcium concentration in unstimulated saliva collected at baseline (before mouthwash(es)), 16, 30, 61, 90 and 121 minutes after mouthwash(es) was expressed as the area under the curve of calcium concentration in saliva as a function of time (millimolar x min).
Time Frame: Baseline, 16, 30, 61, 90 and 121 minutes after a mouthwash(es)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milimolar x minutes
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
Number analyzed (Participants) | 14 | 17
milimolar x minutes | 176 (46.5) | 242 (63.8)
Statistical Analysis 1: Comparison: Fluoride Mouthwash vs Calcium Mouthwash Before Fluoride Mouthwash; A paired t-test was used to compare the two groups; Test type: Superiority; p = 0.0004, t-test, 2 sided — The threshold for statistical significance was set at p=0.05; Paired t-test was used; there were 13 pairs of data, DF=12; Mean Difference (Net) = 50.38, 95% CI 2-sided [27.46 to 73.30] — Treatment difference = Calcium mouthwash before fluoride mouthwash - Fluoride mouthwash

ADVERSE EVENTS:
Time Frame: Until 126 minutes after mouthwash(es) use.
Arm/Group | Fluoride Mouthwash | Calcium Mouthwash Before Fluoride Mouthwash
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

LIMITATIONS AND CAVEATS:
The amount of biofilm collected from participants at the different time points was not enough for all the analyses planned in a number of occasions. This accounts for the lack of data for the calcium concentration in the biofilm fluid.

This experiment was conducted during the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT04239872/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT04239872/ICF_001.pdf